CLINICAL TRIAL: NCT03527654
Title: SER Study: Salud, Estrés, y Resilencia (Health, Stress, and Resilience) Among Young Adult Hispanic Immigrants in the U.S.
Brief Title: SER Hispano Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PRO00087792; 1R01MD012249-01 (NIH)
Record Dates: First submitted 2018-04-27; First posted 2018-05-17 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Stress; Acculturation; Health
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hispanic Immigrants
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Surveys, blood and urine collected prospectively over 24 months.

SUMMARY:
Hispanic immigrants to the U.S. are more likely to experience negative health outcomes the longer they live in the U.S. For example, over time Hispanic immigrants engage in riskier behaviors such as substance abuse, violence, and risky sex, and experience more depressive symptoms. The stress associated with the acculturation process, acculturation stress, and resilience at the individual, family, community, and societal levels appear to play important roles in influencing risks. However, little is known about the causal mechanisms linking acculturation stress, resilience, and health outcomes among Hispanic immigrants. Further, little is known about what precise types of stressors (e.g., occupational stress vs. discrimination) and resilience factors (e.g., individual coping vs. family support) have the most important influence on health trajectories of Hispanic immigrants. The proposed longitudinal study (N = 385) will investigate the effects of acculturation stress and resilience on co-occurring substance abuse, intimate partner violence, HIV risk, and depression (i.e., syndemic conditions) and biological stress among young adult Hispanic immigrants in the U.S. More specifically, the proposed project aims to: 1) test theoretical links between the cumulative impact of acculturation stress and resilience on syndemic conditions and biological stress among recent young adult Hispanic immigrants over a two-year period, and 2) identify the specific types of acculturation stressors and resilience factors at the individual, family, community, and societal levels that are most important in predicting syndemic conditions and biological stress among this population over time. Young adult low-income Hispanic immigrant men and women within the first 10 years of immigration will be followed for two years. Biopsychosocial data will be collected from participants at baseline, and then 6 months (FU1), 12 months (FU2), 18 months (FU3), and 24 months later (FU4). Culturally specific measures of acculturation stress and resilience will be used to assess for individual, family, community, and societal risk and protective factors for syndemic conditions. Blood and urine samples will be obtained from participants to measure systemic inflammation (IL 6, IL8, and IL 18) and oxidative stress (F2 isoprostanes), previously validated biomarkers for psychological stress. Various descriptive, univariate and multivariate statistics, including latent growth curve modeling, will be used to address aims 1-2. The findings from this study have the potential to identify risk and protective factors for the decay in heath among Hispanic immigrants. A precise and culturally informed understanding of these phenomena is foundational for designing interventions that can ultimately promote the health and wellbeing of Hispanic immigrants, the largest immigrant group in the U.S. This study also has the potential to lay the theoretical foundation for biopsychosocial health disparities research in other populations.

ELIGIBILITY:
Inclusion Criteria:

1. identifying as Hispanic or Latino,
2. between 18 and 44 years of age,
3. immigrating to the U.S., and
4. residing in the the U.S. for at least 1 year.

Exclusion criteria will include:

1. acute illness (e.g., cold, flu).

Participants do not need to be able to read, as the questions and responses will be read to the participants.

Ages: 18 Years to 44 Years | Sex: All
Age Groups: Adult
Study Population: Male and female Hispanic immigrants participants between the ages of 18 and 44 living in Durham, Wake, and Orange counties.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Change in syndemic conditions, as measured by the AUDIT, DAST, Revised Conflict Tactics Scale, the Partner table and STI History, the PHQ-9, and the GAD-7. | Baseline, 6 months, 12 months, 18 months, 24 months
  The AUDIT (Babor et. al., 2001) measure has 10 items that assess frequency of drinking and alcohol use disorder symptoms. The DAST (Skinner, 1982) measure, has 10 items that measure drug abuse symptoms. The Revised Conflict Tactics Scale (Strauss & Douglas, 2004) has 24 items that assess conflict between partners and intimate partner violence. The Partner Table & STI History (Gonzalez-Guarda et. al., 2011) has 25 items that assess current sexual practices and risk for sexually transmitted infections including HIV. The PHQ-9 (Kroenke et al., 2002) has 9 items that assess severity depression. The GAD-7 (Spitzer et. al., 2006) contains 7 items that assess anxiety for the individual.
Change in biological stress markers | Baseline, 6 months, 12 months, 18 months, 24 months
  The Inflammatory Cytokines lab test, measures systemic inflammation in body fluid samples (blood and Urine) specifically cytokines IL6, IL8 and IL18. The F2 Isoprostanes measures oxidative stress markers in body fluid samples (blood and Urine) within cells.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Gonzalez-Guarda, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke School of Nursing, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Guarda RM, McCabe BE, Nagy GA, Stafford AM, Matos L, Lu M, Felsman I, Rocha-Goldberg P, Cervantes RC. Acculturative Stress, Resilience, and a Syndemic Factor Among Latinx Immigrants. Nurs Res. 2023 Jul-Aug 01;72(4):249-258. doi: 10.1097/NNR.0000000000000655. Epub 2023 Mar 11. PMID 37350696